CLINICAL TRIAL: NCT02768298
Title: A Randomized, Double-blind, Active-controlled Study to Assess the Effect of LCZ696 Compared With Enalapril to Improve Exercise Capacity in Patients With Heart Failure With Reduced Ejection Fraction (HFrEF).
Brief Title: Exercise Capacity Study of LCZ696 vs. Enalapril in Patients With Chronic Heart Failure and Reduced Ejection Fraction.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLCZ696BDE01; 2015-004632-35 (EudraCT Number)
Record Dates: First submitted 2016-05-09; First posted 2016-05-11 (Estimated); Results first posted 2020-10-09 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Chronic Heart Failure With Reduced Ejection Fraction
Keywords: LCZ696; sacubitril/valsartan; VO2peak; heart failure; systolic heart failure; heart failure with reduced ejection fraction; exercise capacity
MeSH Terms: conditions — Heart Failure; Heart Failure, Systolic | interventions — sacubitril and valsartan sodium hydrate drug combination; Enalapril

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LCZ696 (Experimental): LCZ696 100 mg oral twice daily (bid) for 2 weeks followed by LCZ696 200 mg oral bid for 10 weeks.
  Interventions: Drug: LCZ696; Drug: Placebo matching enalapril
- Enalapril (Active Comparator): Enalapril 5 mg oral twice daily (bid) for 2 weeks followed by enalapril 10 mg oral bid for 10 weeks.
  Patients who prior Screening were at a stable daily dose of enalapril above 10 mg per day (or corresponding doses of other ACEI/ARB) started the study at a dose of enalapril 10 mg bid.
  Interventions: Drug: Enalapril; Drug: Placebo matching LCZ696

INTERVENTIONS:
Drug: LCZ696 — LCZ696 100 mg bid for 2 weeks followed by LCZ696 200 mg bid for 10 weeks. Treatment was administered as oral tablets.
  Arms: LCZ696
Drug: Enalapril — Enalapril 5 mg bid for 2 weeks followed by enalapril 10 mg bid for 10 weeks. Treatment was administered as oral tablets.
  Patients who prior Screening were at a stable daily dose of enalapril above 10 mg per day (or corresponding doses of other ACEI/ARB) started the study at a dose of enalapril 10 mg bid.
  Arms: Enalapril
Drug: Placebo matching enalapril — Patients randomized to LCZ696 arm also received placebo matching enalapril (enalapril 0 mg tablets) to ensure the blinding during the entire course of the study.
  Arms: LCZ696
Drug: Placebo matching LCZ696 — Patients randomized to enalapril arm also received placebo matching LCZ696 (LCZ696 0 mg tablets) to ensure the blinding during the entire course of the study.
  Arms: Enalapril

SUMMARY:
The purpose of the study was to determine the effect of LCZ696 vs. enalapril on improvement of exercise capacity in patients with chronic heart failure with reduced ejection fraction.

DETAILED DESCRIPTION:
This study was a randomized, double-blind, double-dummy, parallel-group, active-controlled, two-arm trial to compare LCZ696 200 mg twice daily (bid) to enalapril 10 mg bid in improving exercise capacity, daily physical activity and quality of life in patients with stable chronic heart failure (New York Heart Association III) and reduced left ventricular ejection fraction (LVEF ≤ 40%).

The study consisted of a screening period of 2 weeks during which the subject's eligibility for the study was assessed followed by a double blind treatment period of 12 weeks. Eligible subjects were randomized 1:1 to receive either LCZ696 or enalapril during the double-blind period. Treatment was initiated with LCZ696 100 mg bid or enalapril 5 mg bid (enalapril 10 mg bid for patients at a stable daily dose of enalapril above 10 mg per day or corresponding doses of other angiotensin converting enzyme inhibitors (ACEI) or angiotensin receptor blockers (ARB) prior first screening visit), respectively. Dose was up-titrated after 2 weeks to the final dose of LCZ696 200 mg bid or enalapril 10 mg bid.

Patients continued to take their background medications for chronic heart failure during the study, with the exception of ACEI or ARBs which were replaced by investigational treatment and had to be discontinued before first dose of study drug.

The primary objective was to demonstrate the superiority of LCZ696 200 mg bid compared to enalapril 10 mg bid in improving exercise tolerance (peak respiratory oxygen uptake (VO2peak), adjusted to body weight) as assessed by cardio-pulmonary-exercise testing (CPET) in patients with stable chronic heart failure (NYHA III) and reduced ejection fraction (LVEF ≤ 40%) after 3 months treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of chronic heart failure (NYHA class III) and reduced ejection fraction (LVEF ≤ 40%)
* Reduced ability to exercise, evidenced by VO2peak ≤ 18 ml/min per kg
* Patients had to be on an ACEI or an ARB at a stable dose of at least enalapril 10 mg/d or equivalent for at least 4 weeks prior to the screening visit and until randomization visit.

Exclusion Criteria:

* History of hypersensitivity or allergy to any of the study drugs, drugs of similar chemical classes, ACEIs, ARBs, or NEP inhibitors as well as known or suspected contraindications to the study drugs
* Previous history of intolerance to recommended target doses of ACEIs or ARBs
* Known history of angioedema
* Requirement of treatment with both ACEIs and ARBs
* Current acute decompensated HF (exacerbation of chronic HF manifested by signs and symptoms that may require intravenous therapy)
* Symptomatic hypotension
* Impaired renal function
* Pregnant or nursing (lactating) women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2016-07-12 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- Germany (29):
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Erfurt
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Koblenz
  - Novartis Investigative Site, Koeln-Nippes
  - Novartis Investigative Site, Leverkusen
  - Novartis Investigative Site, Ludwigsburg
  - Novartis Investigative Site, Ludwigshafen
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Neuwied
  - Novartis Investigative Site, Nienburg
  - Novartis Investigative Site, Rotenburg an der Fulda
  - Novartis Investigative Site, Rüdersdorf
  - Novartis Investigative Site, Siegen
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Villingen-Schwenningen
  - Novartis Investigative Site, Worms
  - Novartis Investigative Site, Wuppertal
  - Novartis Investigative Site, Würzburg

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=647

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 34 investigative sites in Germany.
Pre-assignment Details: Participants were randomized 1:1 to receive either LCZ696 or enalapril during the double-blind period.
Period: Overall Study
Arm/Group | LCZ696 | Enalapril
Started | 103 | 98
Completed | 99 | 91
Not Completed | 4 | 7
Not completed — Adverse Event | 1 | 4
Not completed — Death | 2 | 1
Not completed — Non-compliance with study treatment | 0 | 1
Not completed — Subject/guardian decision | 1 | 0
Not completed — Withdrawal of informed consent | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LCZ696 | Enalapril | Total
Number analyzed (Participants) | 103 | 98 | 201
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.1 (10.792) | 67.6 (9.961) | 66.9 (10.396)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 21 | 38
  Male | 86 | 77 | 163
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucassian | 101 | 96 | 197
  Black | 0 | 1 | 1
  Other | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Peak Respiratory Oxygen Uptake (VO2peak) Adjusted to Body Weight) After 3 Months of Treatment
Description: Cardiopulmonary exercise testing (CPET) is an established method to evaluate the exercise tolerance of heart failure patients by evaluating the cardio-pulmonary system using the measurement of respiratory gases during physical (exercise) stress. One of the parameters attained by this test is the peak respiratory oxygen uptake (VO2peak).
  CPET to assess VO2peak was performed at a cycle ergometer at baseline (Visit 2, 9 days prior randomization) and after 6 weeks and 3 months of treatment (Visit 6 and Visit 7, respectively).
  The VO2peak adjusted to body weight was calculated based on the corresponding visit's VO2peak (unadjusted) and body weight data by using the following formula: VO2peak (unadjusted)/body weight.
  Higher values of VO2peak indicate less symptom severity and therefore a positive change from baseline indicates improvement.
Time Frame: Baseline, 3 months
Population: Full Analysis Set including patients with a valid measurements for the outcome measure.
Measure: Least Squares Mean (Standard Error); unit: mL/kg/min
Arm/Group | LCZ696 | Enalapril
Number analyzed (Participants) | 98 | 90
mL/kg/min | 0.51 (0.180) | 0.19 (0.188)
Statistical Analysis 1: Comparison: LCZ696 vs Enalapril; Test type: Superiority; p = 0.2327, ANCOVA; Least Squares (LS) Mean = 0.32, 95% CI 2-sided [-0.21 to 0.85], Standard Error of Mean 0.268

2. Secondary Outcome: Change From Baseline in Peak Respiratory Oxygen Uptake (VO2peak) Adjusted to Body Weight) After 6 Weeks of Treatment
Description: Cardiopulmonary exercise testing (CPET) is an established method to evaluate the exercise tolerance of heart failure patients by evaluating the cardio-pulmonary system using the measurement of respiratory gases during physical (exercise) stress. One of the parameters attained by this test is the peak respiratory oxygen uptake (VO2peak).
  CPET to assess VO2peak was performed at a cycle ergometer at baseline (Visit 2, 9 days prior randomization) and after 6 weeks and 3 months of treatment (Visit 6 and Visit 7, respectively).
  The VO2peak adjusted to body weight was calculated based on the corresponding visit's VO2peak (unadjusted) and body weight data by using the following formula: VO2peak (unadjusted)/body weight.
  A positive change from baseline indicates less symptom severity.
Time Frame: Baseline, 6 weeks
Population: Full Analysis Set including patients with a valid measurements for the outcome measure.
Measure: Least Squares Mean (Standard Error); unit: mL/kg/min
Arm/Group | LCZ696 | Enalapril
Number analyzed (Participants) | 97 | 88
mL/kg/min | 0.28 (0.185) | 0.42 (0.195)
Statistical Analysis 1: Comparison: LCZ696 vs Enalapril; Test type: Superiority; p = 0.6247, ANCOVA; LS Mean = -0.14, 95% CI 2-sided [-0.68 to 0.41], Standard Error of Mean 0.277

3. Secondary Outcome: Change From Baseline in the Minute Ventilation (VE) to Carbon Dioxide Output Slope (VE/VCO2 Slope)
Description: Cardiopulmonary exercise testing (CPET) is an established method to evaluate the exercise tolerance of heart failure patients by evaluating the cardio-pulmonary system using the measurement of respiratory gases during physical (exercise) stress. One of the parameters attained by this test is the minute ventilation (VE) to carbon dioxide output slope (VE/VCO2 slope). High values of VE/VCO2 slope resembles the inability to eliminate CO2 by respiration (inefficient ventilation).
  A negative change from baseline indicates less symptom severity.
Time Frame: Baseline, 6 weeks, 3 months
Population: Full Analysis Set including patients with a valid measurements for the outcome measure.
Measure: Least Squares Mean (Standard Error); unit: no units
Arm/Group | LCZ696 | Enalapril
Number analyzed (Participants) | 103 | 98
no units
  6 weeks: number analyzed (Participants) | 96 | 87
  6 weeks | -1.05 (0.597) | 0.18 (0.629)
  3 months: number analyzed (Participants) | 93 | 83
  3 months | 0.76 (0.542) | -0.07 (0.575)
Statistical Analysis 1: Comparison: LCZ696 vs Enalapril; 6 weeks; Test type: Superiority; p = 0.1678, ANCOVA; LS Mean = -1.23, 95% CI 2-sided [-2.98 to 0.52], Standard Error of Mean 0.888
Statistical Analysis 2: Comparison: LCZ696 vs Enalapril; 3 months; Test type: Superiority; p = 0.3052, ANCOVA; LS Mean = 0.83, 95% CI 2-sided [-0.77 to 2.43], Standard Error of Mean 0.809

4. Secondary Outcome: Change From Baseline in Exercise Capacity (Watt) at Ventilatory Anaerobic Threshold (VAT)
Description: Cardiopulmonary exercise testing (CPET) is an established method to evaluate the exercise tolerance of heart failure patients by evaluating the cardio-pulmonary system using the measurement of respiratory gases during physical (exercise) stress. CPET was performed at a cycle ergometer with a workload that started at 10 watts (W) and then increased by 10W for each 1-minute stage.
  Exercise capacity assessed as workload in watts was determined at the ventilatory anaerobic threshold (VAT) which represents the transition from aerobic to partially anaerobic glucose metabolism in muscle, leading to increasing carbon dioxide exhalation in comparison to oxygen uptake.
  A positive change from baseline in exercise capacity (watt) indicates improvement.
Time Frame: Baseline, 6 weeks, 3 months
Population: Full Analysis Set including patients with a valid measurements for the outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Watt
Arm/Group | LCZ696 | Enalapril
Number analyzed (Participants) | 103 | 98
Watt
  6 weeks: number analyzed (Participants) | 91 | 82
  6 weeks | 1.71 (1.168) | 0.83 (1.234)
  3 months: number analyzed (Participants) | 84 | 79
  3 months | 2.45 (1.436) | -0.83 (1.483)
Statistical Analysis 1: Comparison: LCZ696 vs Enalapril; 6 weeks; Test type: Superiority; p = 0.6181, ANCOVA; LS Mean = 0.87, 95% CI 2-sided [-2.58 to 4.32], Standard Error of Mean 1.744
Statistical Analysis 2: Comparison: LCZ696 vs Enalapril; 3 months; Test type: Superiority; p = 0.1254, ANCOVA; LS Mean = 3.28, 95% CI 2-sided [-0.93 to 7.48], Standard Error of Mean 2.124

5. Secondary Outcome: Change From Baseline in Rate of Perceived Exertion (Perceived Dyspnea and Perceived Fatigue) During Exercise Assessed by Borg Scale
Description: The individually perceived exertion, in terms of perceived dyspnea and perceived fatigue, during cardiopulmonary exercise testing (CPET) was assessed by Borg scale which is a 15 point scale, starting from 6 which indicates "No exertion at all" to 20 which means "Maximal exertion".
  Change in Borg scale for both perceived dyspnea and perceived fatigue were measured at different time points at Baseline (Visit 2, 9 days prior randomization) and 3 months of treatment (Visit 7). Maximum value among the time points at every visit was used for the analysis.
  A negative change from baseline in Borg value of perceived dyspnea and perceived fatigue indicates improvement.
Time Frame: Baseline, 3 months
Population: Full Analysis Set including patients with a valid measurements for the outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | LCZ696 | Enalapril
Number analyzed (Participants) | 103 | 98
Score on scale
  Borg value perceived dyspnea: number analyzed (Participants) | 93 | 85
  Borg value perceived dyspnea | -0.19 (0.212) | 0.11 (0.223)
  Borg value perceived fatigue: number analyzed (Participants) | 96 | 85
  Borg value perceived fatigue | -0.04 (0.167) | -0.20 (0.178)
Statistical Analysis 1: Comparison: LCZ696 vs Enalapril; Borg value dyspnea; Test type: Superiority; p = 0.3432, ANCOVA; LS Mean = -0.30, 95% CI 2-sided [-0.93 to 0.33], Standard Error of Mean 0.317
Statistical Analysis 2: Comparison: LCZ696 vs Enalapril; Borg value fatigue; Test type: Superiority; p = 0.5319, ANCOVA; LS Mean = 0.16, 95% CI 2-sided [-0.34 to 0.65], Standard Error of Mean 0.251

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 30 days (16 weeks on average).
Description: Any signs or symptoms that occurs during study treatment plus the 30 days post treatment.
Arm/Group | LCZ696 | Enalapril
All-Cause Mortality (participants affected / at risk) | 2/103 | 1/98
Serious Adverse Events (participants affected / at risk) | 12/103 | 14/98
Other Adverse Events (participants affected / at risk) | 52/103 | 36/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 (N=103) | Enalapril (N=98)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Aortic valve incompetence (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Atrial tachycardia (Cardiac disorders) | 0 | 1
Atrial thrombosis (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 2
Cardiogenic shock (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Vascular stent occlusion (General disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Gastroenteritis norovirus (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Septic shock (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Angiocardiogram (Investigations) | 0 | 1
International normalised ratio abnormal (Investigations) | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 2
Renal failure (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 (N=103) | Enalapril (N=98)
Fatigue (General disorders) | 2 | 7
Nasopharyngitis (Infections and infestations) | 9 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 9 | 3
Dizziness (Nervous system disorders) | 14 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Hypotension (Vascular disorders) | 27 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-07-24): https://cdn.clinicaltrials.gov/large-docs/98/NCT02768298/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-10): https://cdn.clinicaltrials.gov/large-docs/98/NCT02768298/SAP_001.pdf